CLINICAL TRIAL: NCT01263522
Title: Optimization of Preventive Effects of Physical Training "Saarländische Ausdauer-Etappe (SAusE)"
Brief Title: Optimization of Preventive Effects of Physical Training
Acronym: SAusE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAusE2011
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Primary Prevention, Cardiovascular Risk Factor Management, Size of Response to Training
Keywords: primary prevention; endurance; cardiovascular risk factors; training; exercise; non-responder
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Endurance training (Experimental)
  Interventions: Other: different training programs
- interval training (Experimental)
  Interventions: Other: different training programs
- strength endurance training (Experimental)
  Interventions: Other: different training programs
- control (Placebo Comparator)
  Interventions: Other: control condition

INTERVENTIONS:
Other: different training programs — two different endurance programs and one strength endurance program
  Arms: Endurance training; interval training; strength endurance training
Other: control condition — unchanged lifestyle
  Arms: control

SUMMARY:
Health-promoting effects of physical exercise are well-investigated especially for endurance activities. However, for different individuals, positive effects have different sizes, even non-responders are observed. Other forms of training, such as strength training and interval training, are less well investigated. Therefore, a comparative longitudinal training study is warranted to examine differences of preventive effects (outcome measures: ergometric descriptors of physical performance, established risk factors and prognostic factors for cardiovascular diseases) of continuous endurance training, interval training and strength endurance training.

In a second stage, the observed non-responders will perform a different type of training (cross-over). It is expected, that besides a comparative general efficacy evaluation of the three training types, improved recommendations for optimized individualization of training parameters can be formulated.

ELIGIBILITY:
Inclusion Criteria:

* untrained
* healthy
* non-smoking

Exclusion Criteria:

* Contraindications for physical activity
* BMI > 30 kg/m2
* resting blood pressure > 160/100 mmHg
* diabetes
* total cholesterol > 300 mg/dl
* maximal oxygen uptake > 50 ml/min/kg for men and > 45 ml/min/kg for women respectively
* other complaints or diseases that might interfere with exercise training

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 266 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
VO2 max | 6 months
  determined during treadmill testing

SECONDARY OUTCOMES:
resting heart rate | 6 months
resting blood pressure | 6 months
blood lipid profile | 6 months
  ratio: total cholesterol/HDL-cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports and Preventive Medicine, Saarland University, Bldg. B 8-2, 66123 Saarbrücken, Saarbrücken, Saarland, Germany

REFERENCES:
- [Derived] Wegmann M, Hecksteden A, Poppendieck W, Steffen A, Kraushaar J, Morsch A, Meyer T. Postexercise Hypotension as a Predictor for Long-Term Training-Induced Blood Pressure Reduction: A Large-Scale Randomized Controlled Trial. Clin J Sport Med. 2018 Nov;28(6):509-515. doi: 10.1097/JSM.0000000000000475. PMID 29189337
- [Derived] Scharhag-Rosenberger F, Meyer T, Wegmann M, Ruppenthal S, Kaestner L, Morsch A, Hecksteden A. Irisin does not mediate resistance training-induced alterations in resting metabolic rate. Med Sci Sports Exerc. 2014 Sep;46(9):1736-43. doi: 10.1249/MSS.0000000000000286. PMID 24566753
- [Derived] Hecksteden A, Wegmann M, Steffen A, Kraushaar J, Morsch A, Ruppenthal S, Kaestner L, Meyer T. Irisin and exercise training in humans - results from a randomized controlled training trial. BMC Med. 2013 Nov 5;11:235. doi: 10.1186/1741-7015-11-235. PMID 24191966